CLINICAL TRIAL: NCT03663478
Title: Ultrasound-guided Transmuscular Quadratus Lumborum Catheters for Elective Caesarean Section. A Double Blind, Randomise, Placebo Controlled Trial.
Brief Title: Continuous TQL Block for Elective Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQL Catheters
Record Dates: First submitted 2018-09-04; First posted 2018-09-10 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Postoperative Pain; Anesthesia, Local
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Ropivacaine
  Interventions: Drug: Ropivacaine
- Control (Placebo Comparator): Isotonic saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ropivacaine — 2 x 30 ml ropivacaine 0,2% and an elastomere pump with 200 ml ropivacaine 0,2%, infusion rate 8 ml/hour
  Arms: Intervention
Drug: Saline — 2 x 30 mL isotonic saline and an elastomere pump with 200 ml isotonic saline, infusion rate 8 ml/hour
  Arms: Control

SUMMARY:
The aim of this study is to investigate whether it is possible to prolong time to first opioid with the TQL block by inserting catheters bilaterally, providing continuous analgesia, in patients undergoing elective CS. Our hypothesis is that it will be possible to significantly extend time to first opioid with the blockade by 66.6%, increasing it from a mean of 5.6 hours to a mean of 10 hours.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age.
* Scheduled for elective Caesarean Section in spinal anaesthesia.
* Have received thorough information, verbally and in written, and signed the "Informed Consent" form on participation in the trial.

Exclusion Criteria:

* Inability to cooperate
* Inability to understand Danish
* Allergy to local anaesthetics or opioids
* Excessive daily intake of opioids, according to the discretion of the investigator
* Local infection at the site of injection or systemic infection
* Difficult visualisation of muscular and fascial structures on ultrasound, necessary to correct blockade and catheter placement.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Time to first opioid | 24 hours postoperatively
  The time from catheters placement to the administration of opioids

SECONDARY OUTCOMES:
Pain intensity (NRS 0-10/10) | 24 hours postoperatively
  NRS (numeric rating scale) score in the study period at 3, 6, 9, 12 and 24 hours postoperatively. In addition, NRS score will be recorded electronically on all morphine administrations, since all patients must enter their NRS score on the Patient-Controlled Analgesia (PCA) pump display prior to administration of the PCA boluses. NRS is a pain scale where the patient gives her pain a number from 0-10, where 0 is no pain and 10 is the worst pain imaginable.
Total morphine consumption. | 24 hours
  Morphine consumption at 3, 6, 9, 12 and 24 postoperative hours (data from PCA pump and patient medical record).
Catheter displacement. | 24 hours
  Frequency of displacement of catheters (early displacement evaluated after 2 hours (T2), late displacement evaluated after 24 hours (T24)).
Patient satisfaction with application of the catheters. | 24 hours
  NRS 0-10/10 during placement of catheters
The degree of morphine-related side effects (PONV, itching, fatigue, etc.). | 24 hours
  On a scale from 0-3, where 0 is none, 1 is mild, 2 is moderate and 3 is severe.
Time from operation to ambulation. | 24 hours
  Time from operation to ambulation.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Børglum, MD PhD, Study Chair — Zealand University Hospital, University of Copenhagen
Locations (1):
- Department of anaesthesiology, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Steingrimsdottir GE, Hansen CK, Borglum J. Ultrasound-guided transmuscular quadratus lumborum catheters for elective caesarean section: A protocol for a single-centre, double-blind randomised trial. Acta Anaesthesiol Scand. 2020 Sep;64(8):1218-1223. doi: 10.1111/aas.13601. Epub 2020 Apr 22. PMID 32270474